CLINICAL TRIAL: NCT00518206
Title: A Phase II Study of the Clinical and Immunological Effects of NY-ESO-1 ISCOM® Vaccine in Patients With Measurable Stage III and IV Malignant Melanoma
Brief Title: Study of NY-ESO-1 ISCOMATRIX® in Patients With Measurable Stage III or IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Austin Health (Other Government); Peter MacCallum Cancer Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2002-013; CTN Trial No.: 2007/123; CTN-Protocol# LUD2002-013AMEND
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Melanoma
Keywords: Clinical Trial; Phase 2; Cancer Vaccine; NY-ESO-1 protein, human; ISCOMATRIX, immunological adjuvant; Cyclophosphamide; T-Cells, Regulatory
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Cohort 1 was enrolled first, in which subjects received the NY-ESO-1 ISCOM vaccine. Enrollment then proceeded to Cohort 2, in which subjects received the NY-ESO-1 ISCOM vaccine and low-dose cyclophosphamide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): NY-ESO-1 ISCOM vaccine (100 μg of the NY-ESO-1 protein formulated with 120 μg of ISCOM adjuvant) administered as an intramuscular injection every 4 weeks for 3 doses in every cycle.
  Interventions: Biological: NY-ESO-1 ISCOMATRIX® vaccine
- Cohort 2 (Experimental): Cyclophosphamide (300 mg/m^2) administered as an intravenous injection 1 day prior to each vaccination with NY-ESO-1 ISCOM (100 μg of the NY-ESO-1 protein formulated with 120 μg of ISCOM adjuvant), which was administered as an intramuscular injection every 4 weeks for 3 doses in every cycle.
  Interventions: Biological: NY-ESO-1 ISCOMATRIX® vaccine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: NY-ESO-1 ISCOMATRIX® vaccine — NY-ESO-1 ISCOM vaccine (100 μg of the NY-ESO-1 protein formulated with 120 μg of ISCOM adjuvant) administered as an intramuscular injection every 4 weeks for 3 doses in every cycle.
Drug: Cyclophosphamide — Cyclophosphamide (300 mg/m^2) administered as an intravenous injection 1 day prior to each vaccination with NY-ESO-1 ISCOM (100 μg of the NY-ESO-1 protein formulated with 120 μg of ISCOM adjuvant), which was administered as an intramuscular injection every 4 weeks for 3 doses in every cycle.
  Arms: Cohort 2

SUMMARY:
This was a Phase 2, open-label study of the NY-ESO-1 ISCOMATRIX® (ISCOM) vaccine administered as an intramuscular injection given every 4 weeks to subjects with measurable advanced malignant melanoma. Study objectives included determination of the anticancer activity, cellular and humoral immunogenicity, and safety and tolerability of the NY-ESO-1 ISCOM vaccine administered alone or preceded by a single administration of low-dose cyclophosphamide.

DETAILED DESCRIPTION:
In Cohort 1, 6 subjects were initially vaccinated with the NY-ESO-1 ISCOM vaccine at a dose of 100 µg of the NY-ESO-1 protein + 120 µg of the ISCOM adjuvant. These 6 subjects were monitored for dose-limiting toxicity (DLT) for 7 days after the first vaccination. Upon observation of tolerability (ie, < 2/6 subjects with DLT), enrollment proceeded to a total accrual of approximately 25 subjects. Subjects received 3 vaccinations administered every 4 weeks (ie, weeks 1, 5, and 9) followed by immunological and clinical response evaluations, with clinical responses categorized according to the Response Evaluation Criteria in Solid Tumors (RECIST). In the absence of disease progression, subjects may have received 3 additional vaccinations administered every 4 weeks, followed by additional vaccinations administered every 12 weeks thereafter until development of disease progression or other criteria for discontinuation.

In Cohort 2, subjects received the NY-ESO-1 ISCOM vaccine on the same schedule as described for Cohort 1, but Cohort 2 subjects also received a single intravenous infusion of low-dose cyclophosphamide 1 day prior to each NY-ESO-1 ISCOM vaccination. If responses were observed in 2 of 16 subjects initially treated in Cohort 2, then 9 additional subjects were to be accrued to Cohort 2, for a total potential accrual of 25 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV (metastatic) or unresectable stage III malignant melanoma.
2. Measurable disease using RECIST.
3. No other effective therapy available or appropriate.
4. Expression of NY-ESO-1 or LAGE-1 by immunohistochemistry (IHC) or reverse transcription-polymerase chain reaction (RT-PCR).
5. Expected survival of at least 4 months.
6. Karnofsky performance status of ≥ 70%.
7. Within 3 weeks prior to first administration of study drug, the following laboratory parameters were required to be within the ranges specified:

   * Hemoglobin ≥ 100 g/L
   * Platelets ≥ 100 x 10^9/L
   * International normalized ratio ≤ 2.0
   * Creatinine ≤ 0.2 mmol/L
   * Bilirubin ≤ 30 mmol/L
8. Age ≥ 18 years.
9. Able and willing to give written informed consent.

Exclusion Criteria:

1. Other serious illnesses, eg, serious infections requiring antibiotics, bleeding disorders, or any condition that in the opinion of the Investigator would have interfered with the ability of the patient to complete all study requirements.
2. Other malignancy within last 3 years, except for treated melanoma or non-melanoma skin cancer or cervical cancer in situ.
3. Known immunodeficiency.
4. Known human immunodeficiency virus positivity.
5. Concomitant systemic treatment with corticosteroids, anti-histaminic drugs, or nonsteroidal anti-inflammatory drugs. Specific cyclooxygenase-2 (COX-2) inhibitors, low-dose aspirin for the prevention of an acute cardiovascular event, and topical or inhaled steroids were permitted.
6. Chemotherapy and/or radiotherapy within 4 weeks prior to study week 1.
7. Other immunotherapy within 4 weeks prior to study week 1.
8. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
9. Lack of availability for immunological and clinical follow-up assessment.
10. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
11. Pregnancy or breastfeeding.
12. Women of childbearing potential: refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-11-28 (Actual); Primary Completion 2010-01-22 (Actual); Study Completion 2010-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Cebon, FRACP, MBBS, PhD, Principal Investigator — Ludwig Institute for Cancer Research - Oncology Unit; Ian D Davis, FRACP, FAChPM, MBBS, PhD, Principal Investigator — Ludwig Institute for Cancer Research - Oncology Unit
Locations (2):
- Australia (2):
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Austin Health (Ludwig Institute Oncology Unit), Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Data have been published

REFERENCES:
- [Result] Nicholaou T, Ebert LM, Davis ID, McArthur GA, Jackson H, Dimopoulos N, Tan B, Maraskovsky E, Miloradovic L, Hopkins W, Pan L, Venhaus R, Hoffman EW, Chen W, Cebon J. Regulatory T-cell-mediated attenuation of T-cell responses to the NY-ESO-1 ISCOMATRIX vaccine in patients with advanced malignant melanoma. Clin Cancer Res. 2009 Mar 15;15(6):2166-73. doi: 10.1158/1078-0432.CCR-08-2484. Epub 2009 Mar 10. PMID 19276262
- [Result] Klein O, Davis ID, McArthur GA, Chen L, Haydon A, Parente P, Dimopoulos N, Jackson H, Xiao K, Maraskovsky E, Hopkins W, Stan R, Chen W, Cebon J. Low-dose cyclophosphamide enhances antigen-specific CD4(+) T cell responses to NY-ESO-1/ISCOMATRIX vaccine in patients with advanced melanoma. Cancer Immunol Immunother. 2015 Apr;64(4):507-18. doi: 10.1007/s00262-015-1656-x. Epub 2015 Feb 7. PMID 25662405

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: NY-ESO-1 ISCOM: Subjects received the NY-ESO-1 ISCOM vaccine (100 μg of the NY-ESO-1 protein formulated with 120 μg of ISCOM adjuvant) administered as an intramuscular injection every 4 weeks for 3 doses in every cycle.
- Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM: Subjects received cyclophosphamide (300 mg/m^2) administered as an intravenous injection 1 day prior to each vaccination with NY-ESO-1 ISCOM (100 μg of the NY-ESO-1 protein formulated with 120 μg of ISCOM adjuvant), which was administered as an intramuscular injection every 4 weeks for 3 doses in every cycle.
Period: Overall Study
Arm/Group | Cohort 1: NY-ESO-1 ISCOM | Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM
Started | 27 | 19
Completed | 16 | 13
Not Completed | 11 | 6
Not completed — Disease Progression Requiring Therapy | 6 | 6
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Drug Supply Issue | 1 | 0
Not completed — Reason Unknown | 1 | 0
Not completed — Completion Status Unknown | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: NY-ESO-1 ISCOM | Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM | Total
Number analyzed (Participants) | 27 | 19 | 46
Age, Continuous [Median (Full Range); unit: years] | 61.0 [36 to 86] | 61.0 [38 to 81] | 61.0 [36 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 27 | 19 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 26 | 13 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 6 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 27 | 19 | 46
Karnofsky Performance Status [Count of Participants; unit: Participants] — Karnofsky scores represent the following performance status categories:
  70: Cares for self; unable to carry on normal activity or to do active work. 80: Normal activity with effort; some signs or symptoms of disease. 90: Able to carry on normal activity; minor signs or symptoms of disease. 100: Normal no complaints; no evidence of disease.
  Participants
    70 | 2 | 0 | 2
    80 | 3 | 1 | 4
    90 | 4 | 8 | 12
    100 | 18 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Best Overall Tumor Response
Description: Tumor responses were evaluated using computed tomography and categorized according to RECIST (version 1.0) at baseline, at week 11, between weeks 23 and 25, and every 12 weeks thereafter. Per RECIST, target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions [no evidence of disease]; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 22 months
Population: Subjects with data available from at least 1 post-baseline response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: NY-ESO-1 ISCOM | Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM
Number analyzed (Participants) | 25 | 19
Participants
  Partial response | 1 | 1
  Stable disease | 12 | 4
  Progressive disease | 12 | 14

2. Secondary Outcome: Cellular Immunogenicity of the NY-ESO-1 ISCOM Vaccine
Description: Blood samples were drawn to measure cellular response at pretreatment and weeks 3, 7, 11, between weeks 23 and 25, week 33, and every 12 weeks thereafter. Cellular immunity included an assay for gamma interferon-producing T cells and enumeration of NY-ESO-1b-specific T cells, detected by fluorescent labeled human leukocyte antigen (HLA)-A2 tetramers carrying the NY-ESO-1b peptide, expressed as percent positive staining of CD4+ and CD8+ T cells. Data are presented for CD4+ and CD8+ T-cell responses (not mutually exclusive) that were pre-existing at baseline (BL) or presented at any time post-BL.
Time Frame: Up to 22 months
Population: Subjects with available results from the evaluation of T-cell responses in peripheral blood.
Measure: Number; unit: participants
Arm/Group | Cohort 1: NY-ESO-1 ISCOM | Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM
Number analyzed (Participants) | 25 | 14
participants
  CD4+ T-cell Response at BL and Post-BL | 4 | 3
  New CD4+ T-cell Response Post-BL | 6 | 7
  CD8+ T-cell Response at BL and Post-BL | 12 | 3
  New CD8+ T-cell Response Post-BL | 5 | 1
  No CD4+ or CD8+ T-cell Response | 6 | 3

3. Secondary Outcome: Post-Vaccination Delayed-type Hypersensitivity (DTH) Reactions
Description: NY-ESO-1-specific DTH was measured by intradermal injection with the full-length NY-ESO-1 protein, NY-ESO-1b peptide, and NY-ESO-1 DP4 peptide at pretreatment, week 11, and between week 23 and 25. DTH reactions (eg, local skin irritation) were evaluated 2 days after DTH injections. Data presented are based on injections with the full-length peptide, as these data are considered to be representative of the comprehensive DTH results.
Time Frame: Up to 22 months
Population: Subjects who underwent DTH testing with available DTH reaction evaluation(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: NY-ESO-1 ISCOM | Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM
Number analyzed (Participants) | 25 | 19
Participants
  Reaction at Pretreatment and Week 11 | 2 | 3
  Reaction at Pretreatment and Week 23 | 1 | 0
  Reaction at Pretreatment, No Reaction On Study | 0 | 1
  Reaction at Pretreatment, No On Study DTH Results | 0 | 1
  No Reaction Pretreatment , Reaction at Week 11 | 6 | 4
  No Reaction Pretreatment , Reaction at Week 23 | 0 | 3
  No Reaction Pretreatment or on Study | 16 | 6
  No Reaction Pretreatment, No On Study DTH Results | 0 | 3

4. Secondary Outcome: Humoral Immunogenicity of the NY-ESO-1 ISCOM Vaccine
Description: Blood samples were drawn to measure humoral immunologic response at pretreatment and weeks 3, 7, 11, 33, and every 12 weeks thereafter. Humoral immunity was assessed by measurement of antibodies to NY-ESO-1 by enzyme-linked immunosorbent assay (ELISA). Data are presented according to baseline (BL) NY-ESO-1 antibody positivity and the time to seroconversion, if applicable.
Time Frame: Up to 22 months
Population: Subjects with available measurement of baseline and post-baseline positivity for NY-ESO-1 antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: NY-ESO-1 ISCOM | Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM
Number analyzed (Participants) | 27 | 15
Participants
  NY-ESO-1 (+) at BL and Post-BL | 7 | 2
  NY-ESO-1 (-) at BL, converted to (+) Post-BL | 19 | 8
  NY-ESO-1 (-) at BL and Post-BL | 1 | 5

5. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (version 3.0). Treatment-emergent adverse events (TEAEs) were reported based on clinical laboratory tests, physical examinations, and vital signs from pre-treatment through the study period. Dose-limiting toxicity was defined as any treatment-related grade 4 toxicity or any grade 3 toxicity, excluding grade 3 skin necrosis at the site of the delayed-type hypersensitivity reaction, fever, or asymptomatic hyperglycemia that improved to baseline within 3 weeks of onset.
Time Frame: Up to 22 months
Population: The Safety Analysis Set comprises all subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1: NY-ESO-1 ISCOM | Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM
Number analyzed (Participants) | 27 | 19
participants
  Any TEAE | 27 | 19
  Maximum Grade 3 TEAE | 4 | 9
  Maximum Grade 4 TEAE | 1 | 1
  Treatment-related TEAE | 26 | 19
  Serious TEAE | 5 | 7
  Death | 0 | 0
  TEAE Leading to Discontinuation | 2 | 1
  Dose-limiting Toxicity | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 22 months.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 3.0), seriousness, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per subject at the maximum reported grade.
Arm/Group | Cohort 1: NY-ESO-1 ISCOM | Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/19
Serious Adverse Events (participants affected / at risk) | 5/27 | 7/19
Other Adverse Events (participants affected / at risk) | 27/27 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: NY-ESO-1 ISCOM (N=27) | Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM (N=19)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant breast lump removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bronchopneumonia (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: NY-ESO-1 ISCOM (N=27) | Cohort 2: Cyclophosphamide + NY-ESO-1 ISCOM (N=19)
Axilliary pain (General disorders) | 3 | 0
Chills (General disorders) | 2 | 1
Fatigue (General disorders) | 10 | 13
Influenza like illness (General disorders) | 6 | 1
Injection site erythema (General disorders) | 5 | 1
Injection site pain (General disorders) | 19 | 16
Pyrexia (General disorders) | 3 | 2
Dizziness (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 5 | 0
Lethargy (Nervous system disorders) | 11 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 4 | 13
Vomiting (Gastrointestinal disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Post procedural infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 2 | 1
Lymph node palpable (Investigations) | 3 | 0
Weight decreased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 3
Chest discomfort (General disorders) | 0 | 1
Feeling hot (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 1
Abdominal wall mass (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to muscle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Hemisensory neglect (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Blood creatine increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less